CLINICAL TRIAL: NCT02030327
Title: Analysis of Predictive Parameters by Proteomics for Early Diagnosis of Organ Dysfunction in Multiple Trauma Patients - A Pilot Study
Brief Title: Proteomics in Multiple Trauma to Identify Organ Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Jochen Hinkelbein, Priv.-Doz. Dr. med., Universitätsklinikum Köln
Other Study IDs: 12-236
Record Dates: First submitted 2014-01-02; First posted 2014-01-08 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Multiple Trauma
Keywords: proteomics; multiple trauma; organ dysfunction
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum (blood) and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No trauma: n=5 patients
- trauma without organ dysfunction: n=40 patients
- trauma with organ dysfunction: n=40 patients

SUMMARY:
To analyse differences in protein expression in multiple trauma patients for identification of potential biomarkers to predict organ dysfunction.

DETAILED DESCRIPTION:
The aim of the present study in humans is to analyse differences in protein expression after multiple trauma in patients for identification of potential biomarkers to predict organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* multiple trauma patients
* ISS >16

Exclusion Criteria:

* children
* ISS <16

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: older than 18 years multiple trauma patients ISS >16
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2014-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with disease or death vs. healthy | Day 0 until day 20
  Starting at day O, then every 24 hours until day 20

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hinkelbein, MD, Principal Investigator — UK Köln
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany